CLINICAL TRIAL: NCT04067505
Title: An Efficacy and Safety Study of Rivaroxaban for the Prevention of Deep Vein Thrombosis in Patients With Left Iliac Vein Compression Treated With Stent Implantation (PLICTS)：A Prospective Randomized Controlled Trial
Brief Title: Rivaroxaban for the Prevention of Deep Vein Thrombosis in Patients With Left Iliac Vein Compression - The PLICTS Study
Acronym: PLICTS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Huadong Hospital (Other); Shanghai Zhongshan Hospital (Other); Shanghai 5th People's Hospital (Other); Yantai Yuhuangding Hospital (Other); Anhui Provincial Hospital (Other Government); Zhejiang Provincial People's Hospital (Other); Zhejiang Hospital (Other)
Responsible Party: Principal Investigator, Zhenjie Liu, Principal Investigator, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZhejiangU-001
Record Dates: First submitted 2019-07-24; First posted 2019-08-26 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: May-Thurner Syndrome
Keywords: May-Thurner Syndrome; warfarin; rivaroxaban; stent implantation
MeSH Terms: conditions — May-Thurner Syndrome | interventions — Rivaroxaban; Warfarin; Nadroparin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Experimental): Participants will receive rivaroxaban 15mg twice daily for three weeks, then 20mg oral once daily after operation.
  Interventions: Drug: Rivaroxaban
- Warfarin/Nadroparin (Active Comparator): Participants will receive nadroparin 1mg/kg twice daily (subcutaneous), plus warfarin 3mg oral once daily for 5 days after the operation, later warfarin(oral) at individually titrated doses(0.75mg to 18mg) to achieve a target international normalized ratio (INR) of 2.0 to 3.0, once daily until 6 months.
  Interventions: Drug: Warfarin; Drug: Nadroparin

INTERVENTIONS:
Drug: Rivaroxaban — Dose: 15mg twice daily for three weeks, then 20mg once daily until six months after the operation. Application: oral
  Other Names: Xarelto
  Arms: Rivaroxaban
Drug: Warfarin — Dose: 3mg for 5 days after the operation, later 0.75mg to 18mg depending on INR (2.0-3.0) until 6 months Duration: 6 months Frequency: once daily Application: oral
  Other Names: coumadin
  Arms: Warfarin/Nadroparin
Drug: Nadroparin — Dose: 1mg/kg Duration: 5 days after the operation Frequency: twice daily Application: subcutaneous
  Other Names: Fraxiparin
  Arms: Warfarin/Nadroparin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of rivaroxaban for the prevention of deep vein thrombosis in patients with left iliac vein compression treated with stent implantation.

DETAILED DESCRIPTION:
Left Iliac Vein Compression Syndrome (LIVCS) is a disease of iliac vein stenosis/occlusion caused by chronic friction and compression of the left iliac vein by the right common iliac artery and lumbar vertebra. It is also called Cockett syndrome or May-Thurner syndrome. Recently, left iliac vein balloon dilatation with stent implantation have been used to treat patients with LIVCS, and have achieved good results. However, no matter the iliac vein stenosis or occlusion, interventional therapy can directly cause local trauma and intimal injury, which is a clear inducement of local thrombosis. Therefore, high intensity anticoagulation therapy is still needed to prevent secondary thrombosis in stent after left iliac vein balloon dilatation with stent implantation. At present, the postoperative anticoagulation regimen of these patients is early heparin anticoagulant therapy, and later warfarin anticoagulant therapy. However, due to the narrow therapeutic window of the drug, patients need to adjust the dosage according to coagulation function under the guidance of doctors. Rivaroxaban can simplify treatment, and is safe. Previous studies have shown that rivaroxaban is effective in preventing deep venous thrombosis after orthopaedic surgery. Rivaroxaban has also been shown to be safe and effective in anticoagulation therapy for patients with deep venous thrombosis and pulmonary embolism. However, Rivaroxaban lacks sufficient clinical data for adjuvant anticoagulation therapy after balloon dilatation with stent implantation. Therefore, this study should be carried out to provide the basis for LIVCS treatment guidelines and explore the clinical indications of rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thrombotic left iliac vein compression syndrome who underwent left iliac vein stent implantation

Exclusion Criteria:

* Age < 18 years or age > 75 years
* With history of pelvic surgery, left iliac vein trauma and pelvic radiotherapy
* With obvious contraindications for anticoagulation therapy
* Allergic to iodine contrast agents in the past
* With concomitant diseases that need high-intensity anticoagulation, and the anticoagulation intensity is clearly higher than that of the patients with iliac vein therapy alone
* Active bleeding or potential bleeding risk
* Pregnant or breastfeeding women
* With pelvic tumors causing compression of left iliac vein,
* With chronic venous insufficiency of lower extremities caused by K-T syndrome
* With malignant tumors and life expectancy < 1 year
* Taking cytochrome P450 3A4(CYP-450 3A4) inhibitors or inducers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
stent occlusion rate | 2 year after operation
  Stent occlusion is defined as DS > 50% for each modality with no procedure performed on the treated segment

SECONDARY OUTCOMES:
Quality of Life Change Scale Survey Results | 1, 3, 6, 12, 18 and 24 months after operation
  Quality of life will be assessed by MOS item short-form health survey scale (SF-36). SF-36 includes eight subscales: physical functioning (PF, 10 items), role limitations due to physical health problems (RL-P, 4 items), bodily pain (BP, 2 items), general health (GH, 5 items), vitality (V, 4 items), social functioning (SF, 2 items), role limitations due to emotional problems (RL-E, 3 items) and mental health (MH, 5 items). The vitality sub-score assesses energy and fatigue, and ranges from 0 (worst) - 100 (best).
All cause mortality | 1, 3, 6, 12, 18 and 24 months after operation
  Percentage of participants with all deaths
anticoagulation raleted mortality | 1, 3, 6, 12, 18 and 24 months after operation
  Percentage of participants with anticoagulation raleted deaths
Proportion of participants with stent displacement/fracture | 1, 3, 6, 12, 18 and 24 months after operation
  Events will be assessed based on computed tomography (CT) or X ray
Proportion of participants with hemorrhage | 1, 3, 6, 12, 18 and 24 months after operation
  Including hemorrhagic stroke, gastrointestinal bleeding, hematuria, mucocutaneous hemorrhage and other visceral bleeding
Proportion of participants with other vascular events | 1, 3, 6, 12, 18 and 24 months after operation
  All vascular events (ST segment elevation myocardial infarction, non ST segment elevation myocardial infarction, acute coronary syndrome, unstable angina, ischemic stroke, transient ischemic attack, pulmonary embolism, non-central nervous system systemic embolism or vascular death) will be assessed based results/films/images of confirmatory testing, and/or case summaries.
Proportion of participants with thrombosis | 1, 3, 6, 12, 18 and 24 months after operation

CONTACTS AND LOCATIONS:
Overall Officials: Zhejie Liu, MD,PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (9):
- China (9):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Yantai Yuhuangding Hospital, Yantai, Shangdong
  - Huadong Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai 5th People's Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The second affiliated hospital of zhejiang university school of medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial people's hospital, Hangzhou, Zhejiang
  - Zhejiang Xiaoshan Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Background] Liu Z, Gao N, Shen L, Yang J, Zhu Y, Li Z, Si Y. Endovascular treatment for symptomatic iliac vein compression syndrome: a prospective consecutive series of 48 patients. Ann Vasc Surg. 2014 Apr;28(3):695-704. doi: 10.1016/j.avsg.2013.05.019. Epub 2013 Oct 27. PMID 24559785
- [Background] O'Sullivan GJ, Semba CP, Bittner CA, Kee ST, Razavi MK, Sze DY, Dake MD. Endovascular management of iliac vein compression (May-Thurner) syndrome. J Vasc Interv Radiol. 2000 Jul-Aug;11(7):823-36. doi: 10.1016/s1051-0443(07)61796-5. PMID 10928517
- [Background] Hurst DR, Forauer AR, Bloom JR, Greenfield LJ, Wakefield TW, Williams DM. Diagnosis and endovascular treatment of iliocaval compression syndrome. J Vasc Surg. 2001 Jul;34(1):106-13. doi: 10.1067/mva.2001.114213. PMID 11436082
- [Background] Eriksson BI, Kakkar AK, Turpie AG, Gent M, Bandel TJ, Homering M, Misselwitz F, Lassen MR. Oral rivaroxaban for the prevention of symptomatic venous thromboembolism after elective hip and knee replacement. J Bone Joint Surg Br. 2009 May;91(5):636-44. doi: 10.1302/0301-620X.91B5.21691. PMID 19407299
- [Background] Turpie AG, Lassen MR, Davidson BL, Bauer KA, Gent M, Kwong LM, Cushner FD, Lotke PA, Berkowitz SD, Bandel TJ, Benson A, Misselwitz F, Fisher WD; RECORD4 Investigators. Rivaroxaban versus enoxaparin for thromboprophylaxis after total knee arthroplasty (RECORD4): a randomised trial. Lancet. 2009 May 16;373(9676):1673-80. doi: 10.1016/S0140-6736(09)60734-0. Epub 2009 May 4. PMID 19411100
- [Derived] Li M, Zhang L, Zhang K, Zhu Y, Shi Z, Zhang W, Gao B, Li L, Fang Z, Yin L, Chen B, Liu Z. An efficacy and safety study of rivaroxaban for the prevention of deep vein thrombosis in patients with left iliac vein compression treated with stent implantation (PLICTS): study protocol for a prospective randomized controlled trial. Trials. 2020 Sep 29;21(1):811. doi: 10.1186/s13063-020-04742-z. PMID 32993773